CLINICAL TRIAL: NCT04635878
Title: Study of INFLAmmasomes NLRP3 in Platelets and Leukocytes During SEPSIS in Intensive Care Unit (INFLA-SEPSIS)
Brief Title: INFLAmmasomes NLRP3 in Platelets and Leukocytes During SEPSIS in Intensive Care Unit
Acronym: INFLA-SEPSIS
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/20/0026; 2020-A00593-36 (Other: ID-RCB)
Record Dates: First submitted 2020-11-10; First posted 2020-11-19 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Sepsis
Keywords: NLRP3 inflammasome; platelets; cytokines; thrombus; septic shock; sepsis
MeSH Terms: conditions — Sepsis; Thrombosis; Shock, Septic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be collected in peripheral blood at the admission in intensive care unit, day two, day seven and at discharge to compare inflammasome NLRP3 and others markers during sepsis and after resolution of the disease.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Sepsis group: patients suffering from sepsis hospitalized in intensive care unit
  Interventions: Other: Blood collection
- Control group: patients without infection hospitalized in intensive care unit
  Interventions: Other: Blood collection

INTERVENTIONS:
Other: Blood collection — Blood collection (at admission, two days, one week and at discharge) to analyze the activation of NLRP3 inflammasome in platelets and leukocytes

SUMMARY:
septic shock is the first cause of mortality in intensive care unit. Innate immunity is the body's first line of defense against pathogens

DETAILED DESCRIPTION:
since their discovery, inflammasomes have an important role during inflammatory response following an aggression. There are intracytoplasmic multiprotein complex activated by cellular stress or infections and is responsible for the release of pro-inflammatory cytokines, including IL-1β. One study focused on the role of the NLRP3 inflammasome in monocyte during sepsis has shown its early alteration that is correlated with mortality. Most studies have analysed inflammasomes in nucleated cells, nevertheless, little is known about inflammasomes in platelets. The aim of the study is to analyze the activation of NLRP3 inflammasome in platelets and leukocytes during sepsis, from patients hospitalized in intensive care unit compare to a control group, until its resolution to better understand the pathophysiology of sepsis

ELIGIBILITY:
SEPSIS GROUP:

Inclusion Criteria:

* hospitalized in intensive care unit with central catheter
* age > or = 18 years
* patients suffering from sepsis
* hospitalized from less than72 hours

Exclusion Criteria:

* patients with curatorship or guardianship
* pregnant women
* patients suffering from malignant blood disease
* patients suffering from disease associated with NLRP3 inflammasome activation

CONTROL GROUP:

Inclusion Criteria:

* hospitalized in intensive care unit with central catheter for other reason than infection
* age > or = 18 years

Exclusion Criteria:

* patients with infection disease
* patients with curatorship or guardianship
* pregnant women
* patients suffering from malignant blood disease
* patients suffering from disease associated with NLRP3 inflammasome activation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in intensive care unit in University Hospital of Toulouse
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Activation kinetics of the NLRP3 inflammasome during sepsis until its resolution | From day 0 to the hospital discharge, an average of 1 month
  Activation kinetics of the NLRP3 inflammasome from day 0 to patient discharge measured by the area under curve

SECONDARY OUTCOMES:
Rate of inflammasome NLRP3 activation | Day 0
  Rate of inflammasome NLRP3 activation (measured in blood samples)
Rate of inflammasome NLRP3 activation | Day 2
  Rate of inflammasome NLRP3 activation (measured in blood samples)
Rate of inflammasome NLRP3 activation | Day 7
  Rate of inflammasome NLRP3 activation (measured in blood samples)
Rate of inflammasome NLRP3 activation | Day of hospital discharge, an average of 1 month
  Rate of inflammasome NLRP3 activation (measured in blood samples)
Severity score measured by Sequential Organ Failure Assessment (SOFA) score | Day 0
  Severity score measured by Sequential Organ Failure Assessment (SOFA) score, from 0 to 4; higher score mean worse outcome
Severity score measured by Sequential Organ Failure Assessment (SOFA) score | Day 2
  Severity score measured by Sequential Organ Failure Assessment (SOFA) score, from 0 to 4; higher score mean worse outcome
Severity score measured by Sequential Organ Failure Assessment (SOFA) score | Day 7
  Severity score measured by Sequential Organ Failure Assessment (SOFA) score, from 0 to 4; higher score mean worse outcome
Severity score measured by Sequential Organ Failure Assessment (SOFA) score | Day of hospital discharge, an average of 1 month
  Severity score measured by Sequential Organ Failure Assessment (SOFA) score, from 0 to 4; higher score mean worse outcome
Severity score measured by Simplified Gravity Index 2 | Day 0
  Severity score measured by Simplified Gravity Index 2, score from 0 to 163, higher score mean worse outcome
Severity score measured by Simplified Gravity Index 2 | Day 2
  Severity score measured by Simplified Gravity Index 2, score from 0 to 163, higher score mean worse outcome
Severity score measured by Simplified Gravity Index 2 | Day 7
  Severity score measured by Simplified Gravity Index 2, score from 0 to 163, higher score mean worse outcome
Severity score measured by Simplified Gravity Index 2 | Day of hospital discharge, an average of 1 month
  Severity score measured by Simplified Gravity Index 2, score from 0 to 163, higher score mean worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Fanny BOUNES, PH, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital of Toulouse, Toulouse, France, France

IPD SHARING:
Plan to Share IPD: No